CLINICAL TRIAL: NCT04062903
Title: A Mental Health Social Prescribing Trial (Mind Cymru)
Brief Title: Social Prescribing Improving Mental Health Study
Acronym: SPRING
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID Pandemic
Sponsor: University of South Wales (Other)
Collaborators: MIND Cymru (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRAS260516
Record Dates: First submitted 2019-08-12; First posted 2019-08-20 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Mental Health Wellness 1
Keywords: Waitlist

STUDY DESIGN:
Intervention Model Description: This study will employ a randomised waitlist trial design with mixed methods using a co-productive participatory approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Appointment (Active Comparator): Intervention group who receive the Social Prescription without delay. The effectiveness of the consultation and referral process will be assessed.
  Interventions: Behavioral: Immediate Appointment
- Delayed Appointment (Active Comparator): Waitlist control group who receive social Prescribing after a delay of 20 working days. The effectiveness of the consultation and referral process will be assessed.
  Interventions: Behavioral: Delayed appointment

INTERVENTIONS:
Behavioral: Immediate Appointment — The participant will meet with the MIND Cymru link worker and decide upon a course of action requiring the use of local services appropriate for the participant.
  Arms: Immediate Appointment
Behavioral: Delayed appointment — After a period of delay (Control) The participant will meet with the MIND Cymru link worker and decide upon a course of action requiring the use of local services appropriate for the participant.
  Arms: Delayed Appointment

SUMMARY:
This study aims to evaluate a new social prescribing service delivered by Mind Cymru in four communities in Wales. Mind Cymru have made a new social prescribing service, where a link worker works with a patient who has mild/moderate mental or emotional health problems, to understand their needs and set them goals for the future. The link worker will then help them find a service in their local community that might help them achieve their goals.

The study uses a waitlist trial, which means that some participants will get to meet the link worker and have the intervention straight away, while others will have to wait for 20 working days. From this, the researchers can compare the people who had the intervention straight away with the people who had to wait. Scores on well-being, quality of life and loneliness questionnaires will be used to see the effects of the intervention on patients, whilst information like patient attendance at the General Practioner surgery will be used to see if there is a difference in the patient's use of health services.

DETAILED DESCRIPTION:
This trial will employ a randomised wait-list control design. The study has been co-designed with the research team at University of South Wales, Mind Cymru, the link workers and General Practioners working within the study sites.

The study will assess the effectiveness of services provided through making three sets of comparisons (based on a set of individual- and service-level outcomes over time - comparing between: - The four Local Mind sites (Merthyr and Valleys, Vale of Clwyd, Brecon and District, Ystradgynlais);

* Those who complete the intervention immediately, with those who are in the waitlist group;
* Those who fully complete the social prescribing intervention with those who do not complete or partially the full social prescription but receive care as usual (either because they do not attend or only partially attend); and Participants will be randomly allocated to receive the social prescribing link worker intervention either immediately, or after a waiting period of 20 working days. Participants will be recruited through consultations with healthcare professionals, either their General Practioner, a practice nurse or the Total Nurse Triage system within the doctors surgery. If the healthcare professional identifies that the prospective participant meets the eligibility criteria of the study (experiencing mild/moderate mental health and/or emotional wellbeing disorders, aged 18+ and registered with a General Practioners in Wales), they will provide the prospective participant with an information pack, and ask for permission to contact. If this permission is given they will be subsequently contacted by the link worker at least 2 working days later, to gain verbal consent and for baseline data collection and randomisation.

The study recruitment target is 1,000 participants, randomized into two groups (a control group, n = 500 and an intervention group n = 500). The sample collected across the 3 General Practice clusters over the 24-month period that the study is open. An attrition rate of 5% is expected. Recruitment will end after 18-months, allowing for 6 months to complete the study and follow-up on participants. The service may continue independently of the study.

Data will be collected at a maximum of five time points:

* Prior to randomisation to either the immediate or wait-list arm
* For wait-list controls: in a reminder telephone call at the end of the 20 day wait
* At the end of their intervention with the link worker
* Four weeks after the end of their intervention with the link worker
* Three months after the end of the previous data collection point Data will be collected either over the telephone or during the intervention with the link workers. All link workers who are collecting data will have study specific training for receiving consent and data collection.

The study will take place over a 24-month period, with participant recruitment lasting a total of 18-months. Data analysis will take place at the end of the 24-month period, although transfer of data from the link workers to the research team at University of South Wales will be continuous over the 24-month period. A final report will be produced at the end of the study for the Welsh Government.

ELIGIBILITY:
Inclusion Criteria:

* Primary care service users who are, at the point of referral:
* Experiencing mild/moderate mental health and/or emotional wellbeing disorders (e.g. anxiety or depression)
* Aged 18+ years
* Registered with a General Practioner in Wales

Exclusion Criteria:

* Unable to give written, informed consent
* Unable to answer all questions (WEMWBS and EQ-5D) at baseline
* Worsening of mental health condition to the point where more intensive support is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline. The Short Warwick-Edinburgh Mental Well-Being Scale (SWEMWBS) Score | At Baseline, 4 weeks and 3 months after randomisation.
  SWEMWBS is completed by the participants and allows self reflection on mental well-being before and during involvement in health enhancing activities. Each of the 7 statements can be scored 1 to 5, from "none of the time" to "all of the time". A total score is calculated by summing the 7 individual statement scores. The minimum score is 7 and the maximum is 35. The higher score signifies better mental well-being.
Change from Baseline. Recovering Quality of Life questionnaire (ReQol - 20) | At Baseline, 4 weeks and 3 months after randomisation
  The Recovering Quality of Life questionaire is completed by the participants and allows self-reporting on their journey to recovery. There are twenty statements with five answers, and can be scored 0-4. The minimum score is 0 and the maximum is 80, where 0 indicates poorest quality of life and 80 indicates highest quality of life.
Change from Baseline. The UCLA 3-Item Loneliness Scale | At Baseline, 4 weeks and 3 months after randomisation
  The UCLA 3-Item Loneliness Scale is completed by the participants and allows self-reporting of subjective feelings of loneliness and social isolation. There are three statements, with three answers, with "hardly ever", scoring 1 and "often" scoring 3. The minimum score is 3 and the maximum 9. A score of 3-5 is considered "not lonely" and 6-9 "lonely".

CONTACTS AND LOCATIONS:
Overall Officials: Mark Llewellyn, Study Director — University of South Wales
Locations (1):
- CTMUHB, Llantrisant, RCT, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the data